CLINICAL TRIAL: NCT03623984
Title: Molecular-Guided Surgery for Pancreatic and Gastrointestinal Neuroendocrine Cancers
Brief Title: Molecular-Guided Surgery for Pancreatic and GI Neuroendocrine Cancers
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: no partipants
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sushanth Reddy, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001980
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Neuroendocrine Carcinoma of Pancreas; Carcinoid
Keywords: Gallium-DOTATATE (68); Neuroendocrine Tumors; Pancreatic neuroendocrine Tumors; Molecular; Surgery; Carcinoid
MeSH Terms: conditions — Carcinoid Tumor; Neuroendocrine Tumors | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gallium Dotatate (Experimental): All patients in the study will be undergoing both a 68Gallium-DOTATATE scan for tumor localization and planned surgical resection. Both of these maneuvers are clinically indicated and the standard of care in the care of these patients. Following induction of general endotracheal anesthesia (as required for the surgery portion of treatment), the patients will receive an additional injection of 68Gallium-DOTATATE in the operating room itself. A probe that can detect 68Gallium will be used to identify tumors in the OR within the patient's abdominal cavity for targeted resection.
  Interventions: Drug: Gallium Dotatate

INTERVENTIONS:
Drug: Gallium Dotatate — Radioguided Surgery for Pancreatic- Neuroendocrine Cancers
  Other Names: Gallium-DOTATATE (68)

SUMMARY:
The purpose of this study is to see if the use of 68Gallium- positron emission tomography and computer tomography (PET/CT) scans along with NETSPOT® (Advanced Accelerator Applications USA, Inc.) can better define the localization of Neuroendocrine tumors enhancing the surgical removal of Neuroendocrine tumors (NETs).

DETAILED DESCRIPTION:
A challenge during cancer surgery is determining all sites of malignant disease. Accurate tumor localization is of utmost importance as complete resection increases the chance of cure and improves patient outcomes even when cure is not possible. However, finding the primary tumor can be very challenging and, in some cases, impossible. With the recent FDA approval of a PET tracer (Ga-68 DOTATATE) that binds to somatostatin receptors for imaging neuroendocrine tumors (NETs), the investigator's institution has the opportunity to dramatically improve the surgical care for these patients. Therefore, the aim for this study is to develop a molecular image-guided surgery program starting with GI NETs. GI NETs are malignant neoplasms that are increasing in prevalence. NETs cause a variety of debilitating symptoms, and, as a result, contribute substantially to cancer-related morbidity. Since the primary treatment for NET is surgical resection, NETs are an ideal model to launch a comprehensive image-guided surgery program. Many NETs are metastatic at presentation or will develop metastases during their course, and it is difficult to identify all disease visually and through manual palpation. Failure to surgically resect all disease leads to symptoms, metastatic disease, and multiple surgical interventions. Many institutions have recently begun using Ga-68 DOTATATE for PET/CT imaging of NETs, and this same tracer can be used for intra-operative localization of primary NETs as well as metastases. The primary impediment to using Ga-68 DOTATATE for this purpose is the need to develop and validate a high-energy gamma (HEG) probe for detecting NETs during surgery. This study will explore the new PET tracer technology and begin a molecular image-guided surgery program for NETs. This initial paradigm will be used to develop a molecular image guided approach to other cancers. It is expected that this type of program could usher a new era of cancer management at the investigator's institution at its forefront and improve outcomes for study participants.

ELIGIBILITY:
Inclusion Criteria:

1. At least 19 years of age and older
2. Male or female patient with a suspected diagnosis of a gastrointestinal-pancreatic neuroendocrine tumor (localized or metastatic) to undergo surgery for resection
3. Localization of the tumor with a pre-operative 68Gallium-DOTATATE scan
4. In the Investigator's judgement, participant is mentally competent to provide informed consent to participate in the study.
5. ECOG performance status of 0-1
6. Negative urine pregnancy test at screening, if applicable.

Exclusion Criteria:

1. Participants who are pregnant, lactating, or intending to become pregnant during the study
2. Female participants of child-bearing age who refuse a urine pregnancy test
3. Participants who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
4. Participants who have participated in an investigational surgical, drug, or device study within the past 30 days.
5. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
6. Patients whose tumors do not localize on a 68Gallium-DOTATATE scan

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2023-06-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of intraoperative findings to preoperative PET scan findings | From initial PET scan (2-3 weeks) until completion of the surgery
  PET probes will be used to quantify the level of gallium dotatate in the tumor tissue and be compared to the gallium dotatate uptake of the preoperative PET scan.

SECONDARY OUTCOMES:
Determine threshold levels of gallium dotatate uptake in order to determine tumor involvement | From baseline through 12 months
  Using a high energy PET probe the level of gallium uptake will be compared to histopathology analysis of removed specimen

CONTACTS AND LOCATIONS:
Overall Officials: Sushanth Reddy, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Kirklin Clinic, Birmingham, Alabama, United States